CLINICAL TRIAL: NCT03490812
Title: Assessment of Investigational Positron Emission Tomography and Post-Processing Procedures Performed as Add-ons to Standard of Care Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Professor, University of Cincinnati
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RP0689/2013H0280
Record Dates: First submitted 2018-02-22; First posted 2018-04-06 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: PET Imaging
MeSH Terms: interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Prospective population (Experimental)
  Interventions: Diagnostic Test: PET scan
- Retrospective population (Experimental)
  Interventions: Other: Retrospective data analysis

INTERVENTIONS:
Diagnostic Test: PET scan — Investigational PET scan as add-on to standard-of-care scan
  Arms: Prospective population
Other: Retrospective data analysis — Review of pre-existing data from January 1, 2001 through December 5, 2017
  Arms: Retrospective population

SUMMARY:
The goals of this study are to (1) develop and refine PET post-processing acquisition procedures, (2) generate preliminary and comparative imaging data for potential clinical trials, and (3) retrospectively evaluate standard of care PET imaging acquisitions by comparison with investigational PET imaging acquisitions.

DETAILED DESCRIPTION:
The prospective portion of study will utilize investigational PET acquisitions in addition to standard of care PET imaging to develop and optimize PET acquisition post-processing techniques as well as to generate preliminary and comparative data for potential clinical trials. These post-processing techniques include but are not limited to visual inspection of lesions, normal tissue, sentinel nodes and imaging artifacts, semi-quantitative analysis including the use of rating schemes, and using various published methods for image post-processing. The PET methodologies we plan to use as part of this study will allow us to obtain morphological, functional and molecular information. Patients receiving a standard of care PET will be asked by study personnel if they are interested in undergoing additional investigational acquisitions before or after their standard of care imaging. If the patient agrees, he/she will remain on the same PET scanner for up to an additional 30 minutes while more images are obtained. Each patient will be imaged for no longer than 2 hours (standard of care imaging and additional investigational imaging). A routine clinical report will be generated for the clinically indicated PET by a nuclear medicine physician. Once this routine clinical PET scan is dictated and finalized, a study team member will obtain the report via IHIS and manually remove all identifiers. This report is being obtained for comparative purposes. All the data being compared will be coded using a unique study number. The retrospective portion of this study will involve the review of pre-existing data from January 1, 2001 through December 5, 2017. The data to be reviewed/analyzed includes PET imaging data that has been previously collected in the course of standard clinical care. The PET imaging acquisitions obtained from the retrospective review will be utilized as a comparison to the investigational images obtained during the prospective portion of this study. The criteria that will be utilized to determine how the retrospective data will be utilized includes the following parameters: type of imaging study, diagnosis, age in decades, gender, and availability of data in the imaging archive.

ELIGIBILITY:
Prospective Population:

Inclusion Criteria:

* Male and female volunteers greater than or equal to 18 years of age
* Patients receiving a standard of care PET scan at OSU

Exclusion Criteria:

* Participants who are pregnant or lactating
* Prisoners
* Subjects incapable of giving informed written consent

Retrospective Population:

Inclusion Criteria:

* Male and female patients greater than or equal to 18 years of age
* Patients who have previously received a standard of care PET scan at OSU

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
image quality | through study completion, on average 2-5 years
  assessed by blinded readers
artifacts | through study completion, on average 2-5 years
  assessed by blinded readers
lesion detectability | through study completion, on average 2-5 years
  assessed by blinded readers
image noise | through study completion, on average 2-5 years
  assessed region of interest over target tissue and background

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Knopp, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

DOCUMENTS (1):
  • Study Protocol (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT03490812/Prot_000.pdf